CLINICAL TRIAL: NCT05550389
Title: Genetic Overview of Pulmonary Hypertension
Brief Title: Genetics of Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Gazi University (Other)
Collaborators: ADHAD (Unknown)
Responsible Party: Principal Investigator, Serdar Kula, Professor Doctor, Gazi University
Other Study IDs: gazi23.12.2019/276
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Hypertension
Keywords: genetics; pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the developments in recent years, pulmonary arterial hypertension (PAH) is still a disease with high mortality and morbidity. Although studies on genetic background have increased, the pathogenesis of PAH remains complex and unresolved. The most comprehensive data are related to bone morphogenetic protein receptor type 2 (BMPR2), and in recent years, new responsible or candidate genes have been identified, especially by new generation DNA sequencing In this study, it was aimed to determine the genetic background of patients with PAH and to investigate the genetics of secondary PAH not only HPAH.

DETAILED DESCRIPTION:
In our study, changes in BMPR2, SARS2, KRT8, KRT18, SMAD9, CAV1, KCKN3, CPS1, TBX4, ACVRL1, G6PC3, EIF2AK4 and ENG genes will be screened in patients with PAH. In addition to previously reported changes in the relevant genes, previously unreported changes that are likely to be significant according to insilico methods are presented.

Patients' age, gender, mean follow-up time, underlying congenital heart anomalies, 6-minute walk test (6 MWT), proBNP, catheter measurement values (mPAB, m RAB, Rp/Rs, PVR), vasoreactivity test positivity, World health organization functional classification (WHO-FS), cardiac function measurements by echocardiography, treatments they received will be collected retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* mPAB ≥25 mmHg, pulmonary capillary wedge pressure (PCWP) ≤15 mmHg, PVR index (PVRI) ≥3 WU.m2 in right heart catheterization.

Exclusion Criteria:

* Neonatal pulmonary hypertension

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with seconder PAH and HPAH followed up in pulmonary hypertension centers
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Genetics of Pulmonary Hypertension | baseline
  Determining the genetic background of patients with PAH and detecting genetic changes that may predispose to PAH in patients with secondary PAH other than HPAH.

SECONDARY OUTCOMES:
The effects of mutations of Pulmonary Hypertension on disease | baseline
  The effects of the detected mutations on the age of onset of the disease, the course of the disease and the response to treatment will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
there is not enough data in the study yet.

REFERENCES:
- [Background] Deng Z, Morse JH, Slager SL, Cuervo N, Moore KJ, Venetos G, Kalachikov S, Cayanis E, Fischer SG, Barst RJ, Hodge SE, Knowles JA. Familial primary pulmonary hypertension (gene PPH1) is caused by mutations in the bone morphogenetic protein receptor-II gene. Am J Hum Genet. 2000 Sep;67(3):737-44. doi: 10.1086/303059. Epub 2000 Jul 20. PMID 10903931
- [Background] Girerd B, Montani D, Eyries M, Yaici A, Sztrymf B, Coulet F, Sitbon O, Simonneau G, Soubrier F, Humbert M. Absence of influence of gender and BMPR2 mutation type on clinical phenotypes of pulmonary arterial hypertension. Respir Res. 2010 Jun 10;11(1):73. doi: 10.1186/1465-9921-11-73. PMID 20534176
- [Background] Ma L, Roman-Campos D, Austin ED, Eyries M, Sampson KS, Soubrier F, Germain M, Tregouet DA, Borczuk A, Rosenzweig EB, Girerd B, Montani D, Humbert M, Loyd JE, Kass RS, Chung WK. A novel channelopathy in pulmonary arterial hypertension. N Engl J Med. 2013 Jul 25;369(4):351-361. doi: 10.1056/NEJMoa1211097. PMID 23883380
- [Background] Gurney AM, Osipenko ON, MacMillan D, McFarlane KM, Tate RJ, Kempsill FE. Two-pore domain K channel, TASK-1, in pulmonary artery smooth muscle cells. Circ Res. 2003 Nov 14;93(10):957-64. doi: 10.1161/01.RES.0000099883.68414.61. Epub 2003 Oct 9. PMID 14551239
- [Background] Machado RD, Eickelberg O, Elliott CG, Geraci MW, Hanaoka M, Loyd JE, Newman JH, Phillips JA 3rd, Soubrier F, Trembath RC, Chung WK. Genetics and genomics of pulmonary arterial hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S32-S42. doi: 10.1016/j.jacc.2009.04.015. PMID 19555857
- [Derived] Hayvaci Canbeyli F, Secgen K, Ezgu FS, Tacoy G, Unlu S, Arabaci HO, Pektas A, Inci A, Kaya EB, Sinan UY, Kucukoglu MS, Kula S. The Role of Genetics in Congenital Heart Disease-Associated Pulmonary Arterial Hypertension. Pediatr Cardiol. 2026 Feb;47(2):821-829. doi: 10.1007/s00246-025-03847-z. Epub 2025 Apr 4. PMID 40180617